CLINICAL TRIAL: NCT02605057
Title: Dermatopharmacokinetic Trial of LEO 80185 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LP0076-1081
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2018-11

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 80185 gel (Experimental): LEO 80185 gel will be allocated to 7 different test sites on each subject
  Interventions: Drug: LEO 80185 gel
- Dovobet Ointment (Experimental): Dovobet Ointment will be allocated to 7 different test sites on each subject
  Interventions: Drug: Dovobet(r) Ointment

INTERVENTIONS:
Drug: LEO 80185 gel
  Arms: LEO 80185 gel
Drug: Dovobet(r) Ointment
  Arms: Dovobet Ointment

SUMMARY:
Given that LEO 80185 gel takes effect in the upper layer of the skin, it is important to compare and examine the amount of the drug in the upper layer of the skin with that of Dovobet® Ointment. Therefore, a dermatopharmacokinetic study will be conducted in healty adult male volunteers to evaluate pharmacokinetics of LEO 80185 gel and Dovobet® Ointment in the stratum corneum. In this trial, a single application of LEO 80185 gel and Dovobet® ointment will be applied to multiple test sites on the back of healthy Japanese male adults and the trial is designed to compare the amount of each of the active ingredients at steady state or close-to-steady state between LEO 80185 gel and Dovobet® Ointment. The amount of calcipotriol and betamethasone dipropionate in the stratum corneum will be assessed by use of tape stripping.

DETAILED DESCRIPTION:
The study consists of two phases:

The pilot: The first part, known as the pilot study, will include 8 subjects and will evaluate pharmacokinetic profile of LEO 80185 gel and Dovobet® Ointment by measuring the amount of each of the active ingredients in the stratum corneum.

Pivotal: The second part, known as the pivotal study, is designed to compare the amount of each of the active ingredients at steady state or close-to-steady state between LEO 80185 gel and Dovobet® Ointment. The number of subjects in the pivotal study and the number of application sites for study medications will be based on the results of the pilot study.

The number of subjects included in the trial and design of trial is in line with previous type of DPK trials in Japan and the Japanese guideline

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form has been obtained.
2. Healthy Japanese male subjects according to medical history, physical examination, ECG, vital signs and laboratory tests.
3. Aged 20 to 40 years inclusive.
4. Subjects with enough skin area for application of the investigational products.

Exclusion Criteria:

1. Body Mass Index outside the range 18-25 kg/m²
2. History or presence of alcohol or drug abuse.
3. History of allergic reaction to any medications.
4. Subjects with, or with a history of, systemic or cutaneous disease that could in any way confound interpretation of the trial results (e.g. atopic dermatitis, eczema, psoriasis)
5. Known or suspected hypersensitivity to any component of LEO 80185 gel or Dovobet® ointment.
6. Known or suspected hepatic, renal or cardiac disorders.
7. Known or suspected disorders of calcium metabolism associated with hypercalcaemia or albumin-corrected serum calcium above the reference range from the sample taken during screening.
8. Subjects with any of the following skin diseases/skin abnormalities that impede the assessment of the application site (back):

   * eczema/dermatitis or abnormal pigmentation
   * bruises or scars
   * inflammation due to sunburn
   * history and/or presence of skin allergy such as atopic dermatitis
   * history of drug hypersensitivity
   * Signs of skin irritation/disease/disorders/symptoms or blemishes at the planned site of application (e.g. erythema, dryness, roughness, scaling, scars, moles, sunburn)
9. Subjects suspected of infection based on the infection testing results from the sample taken during screening (Hepatitis B surface antigen, HCV antibiody, HIV antigen/antibody, serological test for syphilis).
10. Use of systemic, locally injected or inhaled corticosteroids within 4 weeks of Day 1.
11. Use of vitamin D or calcium supplements, or systemic vitamin D analogues within 4 weeks of Day 1.
12. Use of any medication (systemic or topical) within 2 weeks of Day 1.
13. Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 months of Day 1.
14. Current participation in any other interventional clinical trial.
15. Previously randomised in this clinical trial.
16. Previous or current photo-induced or photo-aggravated disease (e.g. abnormal response to sunlight).
17. Exposure to excessive or chronic ultraviolet radiation (e.g. sunlight, sun lamps, tanning booths or photo-therapy) within 4 weeks of Day 1.
18. In the opinion of the (sub)investigator, participation in the trial is inappropriate.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The amount of calcipotriol in the stratum corneum | 24 hours
  Concentrations will be used to determine steady state
The amount of betamethasone dipropionate in the stratum corneum | 24 hours
  Concentrations will be used to determine steady state

SECONDARY OUTCOMES:
Safety (Number and type of adverse events) | 24 hours
  Number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Masahiko Takeshi, MD, Principal Investigator — Shinanokai Shinanozaka Clinic
Locations (1):
- Shinanokai Shinanozaka Clinic, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en